CLINICAL TRIAL: NCT03139110
Title: Welcoming Patients in Emergency Departments: Impact of the Mediator
Brief Title: Impact of a Mediator for Patient Intake in Emergency Departments
Acronym: MEDIA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0038
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Violent Aggressive Behavior; Mediation
MeSH Terms: conditions — Aggression; Negotiating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients treated in emergency departments without the presence of a mediator.
- Mediation: Patients treated in emergency departments with the presence of a mediator.
  Interventions: Behavioral: Presence of a mediator in the emergency departments

INTERVENTIONS:
Behavioral: Presence of a mediator in the emergency departments — The mediator tasks are :
  * Be available to patients who can solicit him and respond to their requests for information, in particular on the organization of the emergency departments and on waiting times
  * Have a proactive attitude towards patients showing nervousness signs
  * Report patients expressing the will to leave the emergency departments before medical care
  * Manage conflicts between patients / accompanying persons and emergency staff and also between patients.
  Groups: Mediation

SUMMARY:
Violence in the workplace is becoming a serious phenomenon in the contemporary world of work. Hospital staff, like any employee working in contact with the public, is particularly exposed to this violence. In emergency departments, the number of patients treated and their heterogeneity, the problems of communicating with healthcare professionals, and waiting times, favor conflict situations. In the already tense context of the emergencies, the incivilities or violent acts have an impact on the well-being of professionals. In order to prevent these situations of violence, a solution could be to integrate a professional with specific skills into the teams to perform mediation functions between caregivers and patients.

The aim of the study is to evaluate the impact of the presence of a mediator in emergency services on personal (verbal or physical) attacks on professionals (caregivers, doctors, administrative staff).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older.
* Registered at the reception of the emergency department between 8 am and 8 pm, excluding bank holidays.

Exclusion Criteria:

* Patient with psychiatric disorders or impairment of judgment related to the taking of toxic substances.
* Patients requiring medical care in less than 30 minutes (sort code).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population participating in the study is composed of:
  * patients admitted to the emergency department,
  * persons accompanying patients,
  * professionals of the emergency departments (nurses, MD, administrative staff).
Sampling Method: Non-Probability Sample
Enrollment: 2378 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of violence or aggression by patients directed towards emergency staff | During the patient stay in the emergency department, an average of 3 hours, up to 8 hours.
  The violence or aggression will be collected by professionals of the emergency department. They will be classified in 4 levels of gravity.
Incidence of violence or aggression by patients's accompanying persons directed towards emergency staff | During the patient stay in the emergency department, an average of 3 hours, up to 8 hours.
  The violence or aggression will be collected by professionals of the emergency department. They will be classified in 4 levels of gravity.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Pôle Information Médicale, Evaluation, Recherche - Hospices Civils de Lyon, Lyon
  - Service d'urgences médicales et chirurgicales - Hôpital Edouard Herriot - HCL, Lyon
  - Service médical d'accueil des urgences - Hôpital de la Croix Rousse - HCL, Lyon
  - Service d'accueil des urgences - Centre hospitalier Lyon Sud - HCL, Pierre-Bénite

REFERENCES:
- [Derived] Touzet S, Buchet-Poyau K, Denis A, Occelli P, Jacquin L, Potinet V, Sigal A, Delaroche-Gaudin M, Fayard-Gonon F, Tazarourte K, Douplat M. Impact of the presence of a mediator on patient violent or uncivil behaviours in emergency departments: a cluster randomised crossover trial. Eur J Emerg Med. 2024 Jun 1;31(3):201-207. doi: 10.1097/MEJ.0000000000001121. Epub 2024 Feb 7. PMID 38329117
- [Derived] Charrier P, Occelli P, Buchet-Poyau K, Douplat M, Delaroche-Gaudin M, Fayard-Gonon F, Jacquin L, Potinet V, Sigal A, Tazarourte K, Touzet S. Strategies used by emergency care professionals to handle interpersonal difficulties with patients: a qualitative study. BMJ Open. 2021 Feb 8;11(2):e042362. doi: 10.1136/bmjopen-2020-042362. PMID 33558353